CLINICAL TRIAL: NCT05694338
Title: A Descriptive and Comparative Analysis of Frailty in Rural Versus Urban Cancer Patients Undergoing Major Surgical Oncologic Procedures
Brief Title: Frailty in Patients With Gastrointestinal Cancer Who Are Undergoing Major Surgery
Status: Active, not recruiting | Type: Observational
Sponsor: The Guthrie Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 2212-74
Record Dates: First submitted 2023-01-12; First posted 2023-01-23 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Gastrointestinal Cancer
MeSH Terms: conditions — Gastrointestinal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Major surgery for gastrointestinal cancer: Patients with gastrointestinal cancer who are scheduled for major surgery
  Interventions: Other: Frailty survey

INTERVENTIONS:
Other: Frailty survey — Frailty survey using the Clinical Risk Analysis Index (RAI-C).

SUMMARY:
This research is for patients who have gastrointestinal cancer and have a planned major surgery. The purpose of this research is to identify cancer patients who may be at risk for frailty. Frailty is common in older adults and may include symptoms of weight loss, weakness, fatigue, low activity, slow walking and other illnesses. Frailty may increase the risk of problems after major surgery. The study will involve a survey, a blood sample, and a review of medical records.

DETAILED DESCRIPTION:
The goals of the study are to:

* Describe the rate of frailty in surgical cancer patients
* Assess if frailty correlates with problems (adverse outcomes) after major surgery

Participants taking part will be asked to complete a survey to assess frailty before surgery. The frailty survey is referred to as the Clinical Risk Analysis Index (RAI-C).

Participants will have about 10 ml (2 teaspoons) of blood drawn before surgery. Blood tests will include complete blood count (CBC), vitamin A, creatinine, C-Reactive Protein (CRP), DHEA, albumin, and prealbumin.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or older
* histologically proven gastrointestinal malignancy
* referral for elective major surgical procedures at including operations for upper and lower gastrointestinal malignancies and hepato-pancreato-biliary
* referral for neoadjuvant treatment followed by any of the above major surgical procedures

Exclusion Criteria:

* under 18 years
* pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with gastrointestinal cancer who are referred for elective major surgery
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2023-03-13 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Percent of patients considered frail assessed by Clinical Risk Analysis Index (RAI-C) Scores of 21 or higher | pre-operative
  Assess Clinical Risk Analysis Index (RAI-C) Scores in rural patients referred for major abdominal surgeries. Survey values will be added to yield a final RAI-C score between 0 and 81. Percent of patients considered frail will be defined as Clinical Risk Analysis Index (RAI-C) Scores of 21 or higher

SECONDARY OUTCOMES:
Adverse outcomes after major surgery | 30 days post-operative
  Assess adverse outcomes postoperatively and if their is a correlation with the frailty score

CONTACTS AND LOCATIONS:
Overall Officials: Rebekah Macfie, MD, Principal Investigator — The Guthrie Clinic
Locations (2):
- United States (2):
  - Guthrie Medical Group, East Corning, New York
  - Robert Packer Hospital, Sayre, Pennsylvania